CLINICAL TRIAL: NCT03819036
Title: Qualitative Assessment of Emergency Dental Treatments in the Pitie Salpetriere Hospital
Brief Title: Qualitative Assessment of Emergency Dental Treatments
Acronym: URGDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180366; 2018-A02692-53 (Other: ANSM)
Record Dates: First submitted 2019-01-25; First posted 2019-01-28 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Dental Care
Keywords: Dental emergency; Toothache; Tooth pain
MeSH Terms: conditions — Toothache | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Questionnaires for patients requiring dental emergencies care
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Day 0 : Satisfaction questionnaire immediately after consultation Day 1, Day 3 and Day 7 : Telephone follow-up

SUMMARY:
The objective of the study is to evaluate the efficiency of emergency procedures and patient satisfaction within the GHPS (Groupe Hospitalier Pitié Salpêtrière) Dental Emergency Department.

Pain is the main reason of consultation at dental emergency.

The investigators evaluate the pain felt before and after the intervention of the emergency with questionnaires at the day of the consultation (D0), then with phone interviews at D1, D3 and D7.

The investigators also evaluate the quality of the reception and care provided in the GHPS service using a satisfaction questionnaire completed by the patients at D0.

DETAILED DESCRIPTION:
I. Research progress

Two investigators will take turns in the service for the research duration. They will be responsible for informing patients of the research upon their arrival in the service, for the data collection and telephone follow-ups.

The course of the research will take place as follows:

Day of consultation (D0):

1. Patient information on the research when he arrives in the service; explanation of its objectives, its modalities and constraints.
2. Verification of eligibility criteria.
3. Collection of the patient's non-opposition by the dentist during the consultation
4. Consultation according to the usual care. During this procedure, the practitioner performs a medical history and, according to the patient's answers, completes the "General Information Questionnaire". He carries out the emergency care and explains the postoperative consequences.
5. Patient filling in the satisfaction questionnaire immediately after consultation.

   Telephone follow-up (D1, D3, D7):
6. Telephone follow-up by the interviewer and fill in the questionnaire - in case of non-availability of the patient on day 1, the patient will be recalled on day 2 and the extrapolated data on the slope of the curve between D1 and D2
7. Telephone follow-up by the interviewer on the day and filling in the questionnaire - if the patient is not available on day 3, the patient will be recalled on day 4 and the data extrapolated according to the slope of the curve between D1 and D4; if the patient is not available at D4, he will be recalled to D5 and the extrapolated data between D1 and D5.
8. Telephone follow-up on the interviewer's day and fill in the questionnaire in case of non-availability of the patient on day 7, the patient will be recalled to D8 and the data extrapolated according to the slope of the curve between D3 and D8; if the patient is still not available on D8, he will be recalled to D9 and the extrapolated data between D3 and D9.

II.STATISTICAL ASPECTS

II.1. Statistical justification for the sample size

58,921 patients were received in emergency consultation day and night during the year 2017. A sample of 1% of the population concerned will be constituted.

Patients received in day emergencies (44,191 patients in 2017) will be eligible. On average 121 patients are received daily in emergencies of day, about 600 per week (excluding weekend).

According to a previous study in the department, 50% of patients in care could not be included in the study or were lost to follow-up.

This leads to a number of 300 patients per week.

The study will therefore be conduct over 2 weeks, to include 600 patients, ie 1.3% of the population consulting

II.2. Description of statistical methods

A descriptive analysis of the characteristics of the sample will be performed (age, sex, reason for consultation, diagnosis, prior appointment test, average score of anxiety and pain scores on D0, D1, D3, D7, compliance with instructions and making follow-up appointments,), satisfaction rating, appreciation of the quality of medical care, politeness of staff, waiting time, assessment of the quality of the care setting, the information received, the treatment received, and the recommendation of the service to third parties will be made.

An analysis of the evolution of pain and anxiety scores between D0, D1, D3 and D7 will be performed.

Correlations between the type of treatment and the perceived pain as well as the type of treatment and the perceived anxiety will be made.

II.3. Method of taking into account missing or invalid data

Patients unreachable during the telephone follow-up period will be contacted the next day; the pain and anxiety scores will then be extrapolated from the previous data and the new data collected, by calculating the nearest point on the curve connecting these two data. If they are new unreachable, the data will be considered missing. Data from patients with missing data will be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient reachable by telephone during the week following his / her care in the service
* Collection of the non-opposition of the patient for his participation in research
* Good understanding of the French language

Exclusion Criteria:

* Patient with communication difficulties or difficulties in understanding the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Pain scores evolution 24 hours after treatment | Day 1
  The pain is measured by simple digital scale (ENS).
  The patient notes his pain between 0 and 10.
  0 being the lowest pain, 10 being the highest pain.

SECONDARY OUTCOMES:
Pain scores evolution 3 days ans 7 days after treatment | Day 3 and Day 7
  The pain is measured by simple digital scale (ENS).
  The patient notes his pain between 0 and 10.
  0 being the lowest pain, 10 being the highest pain.
Anxiety score evaluation bound to the care | Day 0, Day 1, Day 3 and Day 7
  Anxiety is measured by simple digital scale (ENS) from 0 to 10.
Welcome quality evaluation from hospital staff | The day of the emergency care (Day 0).
  The reception, cleanliness quality and waiting time will be measured by ENS scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOUCHER, PU-PH, Principal Investigator — Assistance Publique Hoptiaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No